CLINICAL TRIAL: NCT05571098
Title: The Effects of Nurse Navigation Program on Symptom Management and Psychosocial Adjustment Applied to Patients With Colorectal Cancer
Brief Title: The Effects of Nurse Navigation Program on Symptom Management and Psychosocial Adjustment in Colorectal Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Zeynep DÜLGER, Research Assistant, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ZDULGER
Record Dates: First submitted 2022-09-24; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Colorectal Cancer; Psycho-Oncology; Nursing
Keywords: Colorectal Cancer; Nurse Navigation Program; Psycho-Oncology; Symptom Management; Psychosocial Adjustment
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The design type was determined as a randomized controlled experimental study with a pretest-posttest control group, with repeated measurements.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Individualized colorectal cancer education, psycho-oncological counseling, and a nurse-managed telephone support hotline were provided to the individuals in the experimental group within the NNP. Data were collected before NNP (once in the first week after chemotherapy), during NNP (once in the second week after chemotherapy, once in the first week after the next chemotherapy), after NNP (once in the second week after the next chemotherapy). The duration of the interventions performed via the WhatsApp application varied between 45-60 minutes between individuals.
  Interventions: Behavioral: individualized colorectal cancer education; Behavioral: psycho-oncological counseling; Behavioral: telephone support hotline service
- No intervention (No Intervention): No intervention was applied to this group.

INTERVENTIONS:
Behavioral: individualized colorectal cancer education — Subjects taught within the scope of individualized colorectal cancer education:
  * Common symptoms and management related to disease and treatment,
  * Importance of nutrition in the treatment process.
  Arms: Experimental
Behavioral: psycho-oncological counseling — Topics discussed within the scope of psycho-oncological counseling:
  * Psychological state (anxiety, depression, etc.),
  * Coping strategies about the process,
  * Presence of fear about the disease and/or treatment,
  * Lifestyle changes/problems,
  * Changes in body image,
  * Family/friendship/work-related concerns,
  * Additional issues, comments he wishes to convey
  Arms: Experimental
Behavioral: telephone support hotline service — Within the scope of the NNP, a telephone support hotline service was provided to the participants, where they could consult at any time about the subject they wanted.
  Arms: Experimental

SUMMARY:
This study was conducted to examine the effect of the nurse navigation program (NNP) applied to patients with colorectal cancer on symptom management and psychosocial adjustment to the disease. The design type was determined as a randomized controlled experimental study with a pretest-posttest control group, with repeated measurements. For this purpose, individuals were divided into two groups as experimental (n=31) and control (n=31) groups. The study was carried out in Istanbul Lütfi Kırdar City Hospital Oncology Clinic between July 2021 and February 2022, after the necessary permissions were obtained. While individualized colorectal cancer education, psycho-oncological counseling and telephone support services were provided to the individuals in the experimental group under the guidance of nurse within the scope of NNP, no intervention was applied to the control group. In the study, data were collected with three different data collection tools: "Information Form", "Nightingale Symptom Assessment Scale (N-SAS)", "Psychosocial Adjustment To Illness Scale (PAIS/PAIS-SR)". Data were collected before NNP (once in the first week after chemotherapy), during NNP (once in the second week after chemotherapy, once in the first week after the next chemotherapy), after NNP (once in the second week after the next chemotherapy). The duration of the interventions performed via the WhatsApp application varied between 45-60 minutes between individuals. The research was completed with a total of 60 individuals, 30 in the experimental group and 30 in the control group. The data obtained in the study were analyzed using the SPSS (Statistical Package for Social Sciences) for Windows 22.0 program.

DETAILED DESCRIPTION:
Cancer is a leading cause of death worldwide, accounting for approximately 10 million deaths or one in six deaths in 2020 (WHO, 2022). According to cancer data published by GLOBOCAN 2020, colorectal cancer is the third most common cancer and the second most common cause of death among all cancer types (GLOBOCAN, 2020). Cancer, the incidence of which is increasing day by day, can cause serious mental problems and psychological effects in the social life of patients, as well as physical difficulties, and this situation negatively affects the course of the disease (Ülger et al, 2014). When the relevant literature is examined for colorectal cancer patients, pain, nausea, vomiting, impaired bowel function, anorexia and delirium are the most common symptoms in colorectal cancer patients (Kocakuşak et al, 2011; El-Shami et al, 2015). Many cancer patients experience psychosocial symptoms in addition to physical symptoms (Ülger et al, 2014). The most common psychosocial symptoms in cancer patients are usually adjustment disorders, depression, anxiety, decreased life satisfaction or loss of self-confidence (Akechi et al, 2001; Ateşci et al, 2003; Seven et al, 2013; Rashid et al, 2021). Since the treatment process of cancer includes a heavy and long process, it is important for patients to receive psycho-social support to protect their mental health and improve their ability to cope with the disease (Ülger et al, 2014). Patient navigation includes the services provided by professionals (navigators) trained in this field to provide education and support to individuals in overcoming the problems they encounter in the health care system, to encourage them to have cancer screenings, and to guide individuals (Dönmez, 2019). When the relevant literature is examined, although there are many studies on the use of navigation programs in cancer patients, no study on symptom management and psychosocial adjustment in individuals diagnosed with colorectal cancer has yet been found (Sussman et al, 2018; Loiselle et al, 2010; Nam et al, 2019; Young et al, 2010; Shum et al, 2014). In this context, the aim of this study is to examine the effect of the nurse navigation program applied to colorectal cancer patients on symptom management and psychosocial adjustment and to contribute to the relevant literature.

ELIGIBILITY:
Inclusion criteria:

* Being 18 years old and over
* Being colorectal cancer patient
* Having the capability to use WhatsApp application by themselves or their relatives
* Having adequate cognitive status
* Applying to the outpatient chemotherapy unit for chemotherapy treatment
* Volunteering to participate in the study

Exclusion criteria:

* Not knowing their own diagnosis
* Not having sufficient cognitive status
* Not being able to use WhatsApp by themselves or their relatives
* Having a communication barrier
* Not undergoing active chemotherapy
* Not volunteering to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-02-24 (Actual)

PRIMARY OUTCOMES:
Nightingale Symptom Assessment Scale (N-SAS) scores should be lower in the NNP applied group than in the non-applied group. | 33 weeks
  Nightingale Symptom Assessment Scale (N-SAS) is a quality of life scale developed by Gülbeyaz Can and Adnan Aydıner which evaluates the severity of symptoms developing in patients with cancer and its treatment. The scale consists of 38 items in total. The scale has three sub-dimensions: Physical Well-being (items 1-4, 6-15, 23-27 and 37), Social Well-being (items 5 and 16-22) and Psychological Well-being (items 28-36 and 38). The scale is in a 5-point Likert type, and the patient's response to the evaluated item is scored as "0" if it is no, "1" if it is very little, "2" if it is a little, "3" if it is quite a lot, and "4" if it is too much. A high score indicates that the level of being affected by the disease/treatment-related problems is high (Can and Aydiner, 2011).
Psychosocial Adjustment to Illness Scale (PAIS-SR) scores should be lower in the NNP applied group than in the non-applied group. | 33 weeks
  Psychosocial Adjustment to Illness Scale (PAIS-SR) is a scale developed in English by Derogatis in 1986, aiming to evaluate psychosocial adjustment to physical illness (Deragotis, 1986). The Turkish validity and reliability study of the PAIS-SR was carried out by Adaylar (1995). The scale, which consists of 46 items, has seven sub-dimensions: compliance with health care, occupational environment, home environment, sexual relations, extended family relations, social environment, and psychosocial pressure. The lowest score that can be obtained from the scale is 0, and the highest score is 138. Scores below 35 in the scale indicate "good psychosocial adjustment", scores between 35 and 51 indicate "moderate psychosocial adjustment", and scores above 51 indicate "poor psychosocial adjustment" (Adaylar, 1995).

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Dülger, Principal Investigator — zeynep.dulger@sbu.edu.tr; Elif Dönmez, Study Director — elif.donmez@sbu.edu.tr
Locations (1):
- University of Health Sciences, Istanbul, Üsküdar, Turkey (Türkiye)

REFERENCES:
- [Background] Ülger E, Alacacıoğlu A, Gülseren AŞ, Zencir G, Demir L, Tarhan MO. Psychosocial Problems in Cancer and The Importance of Psychosocial Oncology. Journal of Dokuz Eylul University Medical Faculty. 2014; 28(2): 85-92.
- [Background] Kocakuşak A, Yaşar MA, Güler N, Görmüş C, Aydın S, Özer E, Benek S, Pamak S. Retrospective Evaluation of Patients Aged 45 Years or Younger Diagnosed with Colorectal Cancer. Med Bull Haseki 2011;49:110-113.
- [Background] El-Shami K, Oeffinger KC, Erb NL, Willis A, Bretsch JK, Pratt-Chapman ML, Cannady RS, Wong SL, Rose J, Barbour AL, Stein KD, Sharpe KB, Brooks DD, Cowens-Alvarado RL. American Cancer Society Colorectal Cancer Survivorship Care Guidelines. CA Cancer J Clin. 2015 Nov-Dec;65(6):428-55. doi: 10.3322/caac.21286. Epub 2015 Sep 8. PMID 26348643
- [Background] Akechi T, Nakano T, Okamura H, Ueda S, Akizuki N, Nakanishi T, Yoshikawa E, Matsuki H, Hirabayashi E, Uchitomi Y. Psychiatric disorders in cancer patients: descriptive analysis of 1721 psychiatric referrals at two Japanese cancer center hospitals. Jpn J Clin Oncol. 2001 May;31(5):188-94. doi: 10.1093/jjco/hye039. PMID 11450992
- [Background] Atesci FC, Oguzhanoglu NK, Baltalarli B, Karadag F, Ozdel O, Karagoz N. [Psychiatric disorders in cancer patients and associated factors]. Turk Psikiyatri Derg. 2003 Summer;14(2):145-52. Turkish. PMID 12844281
- [Background] Seven M, Akyüz A, Sever N, Dinçer Ş. Studying the Physical and Psychological Symptoms of Patients with Cancer. TAF Preventive Medicine Bulletin. 2013; 12(3):219-224.
- [Background] Rashid A, Aqeel M, Malik B, Salim S. The prevalence of psychiatric disorders in breast cancer patients; a cross-sectional study of breast cancer patients experience in Pakistan. Nature-Nurture Journal of Psychology. 2021; 1(1).
- [Background] Dönmez E. Use of Navigation Systems. In: Can G, editors. Oncology nursing. Istanbul: Nobel Medical Bookstore; 2019. p. 1295-1301.
- [Background] Sussman J, Bainbridge D, Whelan TJ, Brazil K, Parpia S, Wiernikowski J, Schiff S, Rodin G, Sergeant M, Howell D. Evaluation of a specialized oncology nursing supportive care intervention in newly diagnosed breast and colorectal cancer patients following surgery: a cluster randomized trial. Support Care Cancer. 2018 May;26(5):1533-1541. doi: 10.1007/s00520-017-3981-4. Epub 2017 Nov 30. PMID 29189967
- [Background] Loiselle CG, Edgar L, Batist G, Lu J, Lauzier S. The impact of a multimedia informational intervention on psychosocial adjustment among individuals with newly diagnosed breast or prostate cancer: a feasibility study. Patient Educ Couns. 2010 Jul;80(1):48-55. doi: 10.1016/j.pec.2009.09.026. Epub 2009 Oct 24. PMID 19854604
- [Background] Nam KH, Kim HY, Kim JH, Kang KN, Na SY, Han BH. Effects of social support and self-efficacy on the psychosocial adjustment of Korean ostomy patients. Int Wound J. 2019 Mar;16 Suppl 1(Suppl 1):13-20. doi: 10.1111/iwj.13038. PMID 30793862
- [Background] Young J, Harrison J, Solomon M, Butow P, Dennis R, Robson D, Auld S. Development and feasibility assessment of telephone-delivered supportive care to improve outcomes for patients with colorectal cancer: pilot study of the CONNECT intervention. Support Care Cancer. 2010 Apr;18(4):461-70. doi: 10.1007/s00520-009-0689-0. Epub 2009 Jul 22. PMID 19626346
- [Background] Shum NF, Lui YL, Law WL, Fong YTD. A nurse-led psycho-education programme for Chinese carers of patients with colorectal cancer. Cancer Nursing Practice. 2014;13(5): 31-39.
- [Background] Can G, Aydiner A. Development and validation of the Nightingale Symptom Assessment Scale (N-SAS) and predictors of the quality of life of the cancer patients in Turkey. Eur J Oncol Nurs. 2011 Feb;15(1):3-11. doi: 10.1016/j.ejon.2009.10.010. Epub 2009 Nov 26. PMID 19944644
- [Background] Derogatis LR. The psychosocial adjustment to illness scale (PAIS). J Psychosom Res. 1986;30(1):77-91. doi: 10.1016/0022-3999(86)90069-3. PMID 3701670
- [Background] Adaylar AM. Attitude, adaptation, perception and self-care orientations of individuals with chronic disease. PhD Thesis. Istanbul: Istanbul University, Institute of Health Sciences; 1995.
- See also: World Health Organization (2020). Cancer. — https://www.who.int/news-room/fact-sheets/detail/cancer
- See also: GLOBOCAN (2020). — https://gco.iarc.fr/today/data/factsheets/populations/900-world-fact-sheets.pdf